CLINICAL TRIAL: NCT06551818
Title: Prospective, Interventional, Exploratory, Four-Arm - Dose Response Study, Comparative, Double-Blind, Randomized, Placebo-Control, Proof of Concept, Safety, Efficacy and In-Use Tolerability Study of Three Different Dosage Formulation of Test Hair Growth Products and Placebo in Patients With Mild to Moderate Androgenic Alopecia (Grade I to III).
Brief Title: A Clinical Study to Assess Safety, Efficacy and In-use Tolerability of Different Dosages of Hair Growth Products in Patients With Mild to Moderate Androgenic Alopecia (Grade I to III).
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Zywie Ventures Privated Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NB240030-ZV
Record Dates: First submitted 2024-08-02; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Androgenic Alopecia
MeSH Terms: conditions — Alopecia | interventions — Liposomes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SesZen-Bio Low Dose 1 (350 mg extract) (Experimental): Mode of Usage: Swallow the capsule whole with a full glass of water without chewing, crushing, or opening it.
  Dosage form: capsule Frequency: One time daily after meal Rout of administration: Oral
  Interventions: Other: SesZen-Bio Low Dose 1 (350 mg extract)
- SesZen-Bio Low Dose 1 (150 mg liposomal) (Experimental): Mode of Usage: Swallow the capsule whole with a full glass of water without chewing, crushing, or opening it.
  Dosage form: capsule Frequency: One time daily after meal Rout of administration: Oral
  Interventions: Other: SesZen-Bio Low Dose 1 (150 mg liposomal)
- SesZen-Bio High Dose 1 (500 mg extract) (Experimental): Mode of Usage: Swallow the capsule whole with a full glass of water without chewing, crushing, or opening it.
  Dosage form: capsule Frequency: One time daily after meal Rout of administration: Oral
  Interventions: Other: SesZen-Bio High Dose 1 (500 mg extract)
- Placebo (Placebo Comparator): Mode of Usage: Swallow the capsule whole with a full glass of water without chewing, crushing, or opening it.
  Dosage form: capsule Frequency: One time daily after meal Rout of administration: Oral
  Interventions: Other: Placebo

INTERVENTIONS:
Other: SesZen-Bio Low Dose 1 (350 mg extract) — Mode of Usage: Swallow the capsule whole with a full glass of water without chewing, crushing, or opening it.
  Dosage form: Capsule Frequency: One time daily after meal Rout of administration: Oral
  Arms: SesZen-Bio Low Dose 1 (350 mg extract)
Other: SesZen-Bio Low Dose 1 (150 mg liposomal) — Mode of Usage: Swallow the capsule whole with a full glass of water without chewing, crushing, or opening it.
  Dosage form: Capsule Frequency: One time daily after meal Rout of administration: Oral
  Arms: SesZen-Bio Low Dose 1 (150 mg liposomal)
Other: SesZen-Bio High Dose 1 (500 mg extract) — Mode of Usage: Swallow the capsule whole with a full glass of water without chewing, crushing, or opening it.
  Dosage form: Capsule Frequency: One time daily after meal Rout of administration: Oral
  Arms: SesZen-Bio High Dose 1 (500 mg extract)
Other: Placebo — Mode of Usage: Swallow the capsule whole with a full glass of water without chewing, crushing, or opening it.
  Dosage form: Capsule Frequency: One time daily after meal Rout of administration: Oral
  Arms: Placebo

SUMMARY:
This is a prospective, interventional, exploratory, four-arm - dose response study, comparative, double-blind, randomized, placebo-control, proof of concept, safety, efficacy and in-use tolerability study of three different dosage formulation of test hair growth products and placebo in patients with mild to moderate Androgenic Alopecia (Grade I to III).

DETAILED DESCRIPTION:
A total of up to 72 patients (18 patients/arm) preferably equal number of male and female will be enrolled to ensure a total of 60 patients (15 patients/ arm) to complete the study.

There will be total of 8 visits during the study. The duration of the study will be 180 days (6 months) from the enrolment.

Visit 01 (Day -04): Screening, Tattoo creation, hair growth measurement. Visit 02(Day 01):Enrolment, hair growth rate measurement, hair length (androgenic affected targeted area and standard area), hair thickness, hair density, scalp condition for keratin measurement, A: T ratio, number of new hairs, number of hair fall from root, hair root strength, general appearance of hair, general appearance of scalp, earlier product perception questionnaire, global pictures of head crown, CBC, Biochemical tests, free testosterone, testosterone, dihydrotestosterone, CRP, Cortisol random, ferritin, urinalysis.

Visit 03 (Day 45): Hair Length (Androgenic Alopecia affected targeted area standard area), hair thickness, hair density, scalp condition for keratin measurement, hair regrowth (AG affected area), number of hair fall from root, number of new hairs (full scalp and normal scalp- tattoo area), hair root strength, general appearance of hair, general appearance of scalp, product perception questionnaire, global pictures of head crown.

Visit 04 (Day 87): Tattoo creation, hair growth measurement Visit 05 (Day 90):Hair growth rate measurement, hair length (Androgenic Alopecia affected targeted area and standard area), hair thickness, hair density, scalp condition for keratin measurement, A: T ratio, hair regrowth (AG affected area), number of new hairs (on full scalp, normal scalp- tattoo area), number of hair fall from root, hair root strength, general appearance of hair, general appearance of scalp, product perception questionnaire, digital photographs of global pictures head crown.

Visit 06 (Day 135):Hair length (Androgenic Alopecia affected targeted area and standard area), hair thickness, hair density, scalp condition for keratin measurement, hair regrowth (AG affected area), number of hair fall from root, number of new hair (on full scalp, normal scalp- tattoo area), hair root strength from root, general appearance of hair, general appearance of scalp, product perception questionnaire, digital photographs of global pictures head crown.

Visit 07 (Day 177): Tattoo creation, hair growth measurement Visit 08 (Day 180): Hair growth rate measurement, hair length (standard area and Androgenic Alopecia affected targeted area), hair thickness, hair density, scalp condition for keratin measurement, A: T Ratio, number of new hair (on full scalp, AG affected area), hair regrowth (AG affected area), number of hair fall from root, hair root strength, general appearance of hair, general appearance of scalp, product perception questionnaire, global pictures of head crown CBC, Biochemical tests, free testosterone, testosterone, dihydrotestosterone, CRP, Cortisol random, ferritin, urinalysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 25 to 45 years and above (both inclusive) at the time of consent.
2. Sex: Males and non-pregnant/non-lactating females (preferably equal number of males and females).
3. Females of childbearing potential must have a self-reported negative urine pregnancy.
4. Patient is in good general health as determined by the Investigator on the basis of medical history.
5. Patients having mild to moderate Androgenic Alopecia (Grade I to III) during clinical study and grade will be evaluated by the dermatologist by using Norwood-Hamilton classification and Ludwig pattern scale for female.
6. Female with 40-50 counts and male with 25 -30 counts of hair fall at screening.
7. Patient is able to remain on stable doses of contraceptive or replacement hormonal therapy, including no therapy, 6 weeks prior to and for the duration of the study.
8. If the patient is of childbearing potential, is practicing and agrees to maintain an established method of birth control (IUD, hormonal implant device/injection, regular use of birth control pills or patch, diaphragm, condoms with spermicide or sponge with spermicidal jelly, cream or foam, partner vasectomy or abstinence). Females will be considered as non-childbearing potential if they are surgically sterile, have been post-menopausal for at least 1 year or have had a tubal ligation.
9. Patients are willing to give written informed consent and are willing to follow the study procedure.
10. Patients who commit not to use any other medicated/ prescription shampoos/hair care products (containing Minoxidil), any other hair growth products or hair colour or dye, other than the test products for the entire duration of the study.
11. Willing to consume test products throughout the study period.
12. Patient is willing and able to follow and allow study staff to performed study test methods.
13. Patient is willing and able to follow the study directions, to participate in the study, returning for all specified visits.
14. Patient must be able to understand and provide written informed consent to participate in the study.

Exclusion Criteria:

1. Patient have history of severe hair fall due to any clinically significant problems like anaemia, thyroid problems.
2. Patient have history of any dermatological condition of the scalp other than hair loss and dandruff.
3. Patient have history of any prior hair growth procedures (e.g. hair transplant or laser).
4. Patient who had taken topical treatment of hair loss for at least 4 weeks.
5. Patient who had taken any systemic treatment for at least 3 months.
6. History of alcohol or drug addiction.
7. Patient having history or resent condition of irritated or visibly inflamed scalp or severe scalp disease.
8. Patient who is currently participating in or planning on starting weight loss program that may result in a significant change in overall body weight.
9. Pregnant or breast feeding or planning to become pregnant during the study period.
10. History of chronic illness which may influence the cutaneous state.
11. Patient have participated any clinical research study related to hair care products.
12. Patient have history of mastectomy for cancer involving removal of lymph nodes within the past year, or treatment of any type of cancer within the last 6 months.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-08-30 (Estimated); Primary Completion 2025-03-02 (Estimated); Study Completion 2025-03-02 (Estimated)

PRIMARY OUTCOMES:
Change in hair thickness by using CASLite Nova (instrumental analysis) | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90, Day 135 and on Day 180
  To assess the effectiveness of the test products in terms of change in hair thickness
Change in hair density by using CASLite Nova (instrumental analysis) | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90, Day 135 and on Day 180
  To assess the effectiveness of the test products in terms of change in hair density
Change in hair growth rate by using CASLite Nova (instrumental analysis) | 04 before Day 01, Day 01, Day 87, Day 90, Day 177 and on Day 180
  To assess the effectiveness of the test products in terms of change in hair growth rate

SECONDARY OUTCOMES:
Change in keratin measurement from hair by using CASLite Nova (instrumental analysis) | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90, Day 135 and on Day 180
  To assess the effectiveness of the test products in terms of change in keratin from Androgenic Alopecia affected targeted area and normal scalp- tattoo area measurement from hair
Change in hair length | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90, Day 135 and on Day 180
  To assess the effectiveness of the test products in terms of change in hair length (AG affected area and standard area) by using CASLite Nova (instrumental analysis) followed by Image pro-analysis (software analysis)
Change in A:T ratio by hair pluck test | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 90 and on Day 180
  To assess the effectiveness of the test products in terms of change in A:T ratio by dermatologist.
Change hair fall from root test by 60 seconds hair combing test | 04 before Day 01, Day 01, Day 87, Day 90, Day 177 and on Day 180
  To assess the effectiveness of the test products in terms of change hair fall by dermatologist.
Change in number of new hairs by using CASLite Nova (instrumental analysis) | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90, Day 135 and on Day 180
  To assess the effectiveness of the test products in terms of change in number of new hairs
Change in hair regrowth by using CASLite Nova (instrumental analysis) | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90, Day 135 and on Day 180
  To assess the effectiveness of the test products in terms of change in hair regrowth from Androgenic Alopecia affected targeted area
Change in hair root strength | Baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90, Day 135 and on Day 180
  To assess the effectiveness of the test products in terms of change in hair root strength by dermatological assessment
Change in general appearance of hair volume | baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90 and on Day 180
  To assess the effectiveness of the test products in terms of change in general appearance of hair volume in which score done as 1= small 3=full
Change in general appearance of hair plasticity | baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90 and on Day 180
  To assess the effectiveness of the test products in terms of change in general appearance of hair plasticity in which score done as 1=waved and 3=average
Change in general appearance of hair density | baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90 and on Day 180
  To assess the effectiveness of the test products in terms of change in general appearance of hair density in which score as 1=thinned and 2=dense
Change in general appearance of hair dryness | baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90 and on Day 180
  To assess the effectiveness of the test products in terms of change in general appearance of hair dryness in which score done as 1=none, and 4=excessive
Change in general appearance of hair shininess | baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90 and on Day 180
  To assess the effectiveness of the test products in terms of change in general appearance of hair shininess in which score done as 1=poor and 3=good
Change in general appearance of hair smoothness | baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90 and on Day 180
  To assess the effectiveness of the test products in terms of change in general appearance of hair smoothness in which score done as 1=poor, and 3=good
Change in general appearance of hair strength | baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90 and on Day 180
  To assess the effectiveness of the test products in terms of change in general appearance of hair strength in which score done as 1=poor, and 3=good
Change in general appearance of hair oiliness | baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90 and on Day 180
  To assess the effectiveness of the test products in terms of change in general appearance of hair oiliness in which score done as 1=none and 4=excessive
Change in general appearance of scalp Itchiness | baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90 and on Day 180
  To assess the effectiveness of the test products in terms of change in general appearance of scalp Itchiness in which score done as 1= none, and 4=excessive
Change in general appearance of scalp redness | baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90 and on Day 180
  To assess the effectiveness of the test products in terms of change in general appearance of scalp redness in which score done as 1= none, and 4=excessive
Change in general appearance of scalp roughness | baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90 and on Day 180
  To assess the effectiveness of the test products in terms of change in general appearance of scalp roughness in which score done as 1= none, and 4=excessive
Change in general appearance of scalp scaliness | baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90 and on Day 180
  To assess the effectiveness of the test products in terms of change in general appearance of scalp scaliness in which score done as 1=none, and 4=excessive
Change in general appearance of scalp dryness | baseline before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90 and on Day 180
  To assess the effectiveness of the test products in terms of change in general appearance of scalp dryness in which score done as none, mild, moderate and excessive
Change in products perception questionnaire | Before usage of the test products on Day 01 and after usage of the test products on Day 45, Day 90, Day 135 and on Day 180
  To evaluate the effectiveness of the test products in terms of change in products perception questionnaire by using 5-point Likert scale in which 1= not at all and 5= to large extent
Change in tensile strength by TESTRONIX tensile tester (instrumental assessment) | Baseline before usage of test product on Day 01 and after usage of test product on Day 180.
  To assess the effectiveness of the test products in terms of change in tensile strength of hairs
Change in nail brittleness | Baseline before usage of test product on Day 01 and after usage of test products and on Day 180
  To evaluate the effect of test products in terms of change in nail brittleness in which score done by 5 liert scale in which 1-not at all and 5- to large extent
Change in CBC- haemoglobin | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in CBC- haemoglobin
Change in CBC- haematocrit | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in CBC- haematocrit
Change in CBC- RBC (Red Blood Corpuscle) | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in CBC- RBC (Red Blood Corpuscle)
Change in CBC-MCH (mean corpuscular hemoglobin) | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in CBC- MCH (mean corpuscular hemoglobin)
Change in CBC- MCV (mean corpuscular volume) | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in CBC- MCV (mean corpuscular volume)
Change in CBC- MCHC (mean corpuscular haemoglobin concentration) | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in CBC- MCHC (mean corpuscular haemoglobin concentration)
Change in CBC- WBC (White Blood Cell) | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in CBC- WBC (White Blood Cell)
Change in Biochemistry- SGOT (serum glutamic oxaloacetic transaminase) | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in Biochemistry- SGOT (serum glutamic oxaloacetic transaminase)
Change in Biochemistry- SGPT (serum glutamic oxaloacetic transaminase ) | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in Biochemistry- SGPT (serum glutamic oxaloacetic transaminase)
Change in Biochemistry- serum creatinine | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in Biochemistry- serum creatinine
Change in Biochemistry- BUN (blood urea nitrogen) | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in Biochemistry- BUN (blood urea nitrogen)
Change in Biochemistry- RBS (random blood sugar) | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in Biochemistry- RBS (random blood sugar)
Change in Biochemistry- PPBS (post-prandial blood sugar) | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in Biochemistry- PPBS (post-prandial blood sugar)
Change in Biochemistry- TC (Total cholesterol ) | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in Biochemistry- TC (Total cholesterol )
Change in Biochemistry- TG (Triglyceride levels) | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in Biochemistry- TG (Triglyceride levels)
Change in Biochemistry- HDL (high-density lipoproteins) | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in Biochemistry- HDL (high-density lipoproteins)
Change in Biochemistry- LDL (low-density lipoproteins) | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in Biochemistry- LDL (low-density lipoproteins)
Change in Biochemistry- uric acid | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in Biochemistry- uric acid
Change in Biochemistry- VLDL (very low-density lipoprotein) | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in Biochemistry- VLDL (very low-density lipoprotein)
Change in testosterone | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in testosterone
Change in free testosterone | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in free testosterone
Change in dihydrotestosterone | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in dihydrotestosterone
Change in CRP (C-reactive protein) | Before usage of test products on Day 01 from baseline and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in CRP (C-reactive protein)
Change in random cortisol | Before usage of test products on Day 01 from baseline and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change random cortisol
Change in ferritin | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in ferritin
Change in urinalysis - albumin | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in urinalysis-albumin
Change in urinalysis-blood | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in urinalysis-blood
Change in urinalysis-glucose | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in urinalysis-glucose
Change in urinalysis-pH | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in urinalysis-pH
Change in urinalysis-colour | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in urinalysis-colour
Change in urinalysis-appearance | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in urinalysis-appearance
Change in urinalysis-deposits | Baseline before usage of test products on Day 01 and after usage of test products on Day 180
  To evaluate the effect of test products in terms of change in urinalysis-deposits

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nayan K Patel, Principal Investigator — NovoBliss Research Pvt Ltd

IPD SHARING:
Plan to Share IPD: No